CLINICAL TRIAL: NCT03715985
Title: A Pilot Study of the Safety, Tolerability, Feasibility and Efficacy of Anti-PD-1 or Anti-PD-L1 in Combination With a Personalized Neo-antigen Vaccine in Advanced Solid Tumors (NeoPepVac)
Brief Title: Personalized Neo-antigen Vaccine in Advanced Solid Tumors (NeoPepVac)
Acronym: NeoPepVac
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Inge Marie Svane, Clinical Professor, Herlev Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AA1833
Record Dates: First submitted 2018-10-17; First posted 2018-10-23 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Malignant Melanoma, Metastatic; Non Small Cell Lung Cancer Metastatic; Bladder Urothelial Carcinoma, Metastatic
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Not a randomized study. 25 patients to be included. Group A) has not yet started standard treatment Group B) has begun standard treatment at least 4 months before first vaccine, and the decease development is status quo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoPepVac (Experimental): Group A (has not yet started standard treatment) and Group B (has begun standard treatment at least 4 months before first vaccine, and the decease development is status quo) will receive 6 vaccines in total. Firstly 3 vaccines intraperitoneal biweekly and lastly 3 vaccines intramuscular biweekly while the patients are receiving standard immune therapy.
  Interventions: Drug: EVAX-01-CAF09b

INTERVENTIONS:
Drug: EVAX-01-CAF09b — The personalised NPV-ds001 drug substance consists of multiple linear peptides (Pep-Ints) comprising natural L-amino acids dissolved in Dimethyl sulfoxide (DMSO) and 1 ml adjuvants (CAF09b) and 1,08 ml Tris buffer (25 ml).
  Other Names: NPV-ds001-CAF09b

SUMMARY:
The primary objective is to assess tolerability and safety of a personalized neo-antigen vaccine containing up to 15 peptides derived from somatic mutation of the individual patient's cancer, with CAF09b as adjuvant. The vaccine formulation will be administered in combination with an approved anti-PD-1 or anti-PD-L1 inhibitor to patients with advanced solid tumors. The endpoint is the characterization of adverse events (AE) assessed by CTCAE 4.0.

The secondary objective is feasibility to manufacture a personalized neo-antigen vaccine within 6 weeks of enrolment with the PIONEER pipeline, and to evaluate the immune response before, during and after treatment with the personalized neo-antigen vaccine. And evaluate the effect on the immune response correlated to dose escalation of peptides in the vaccine. The endpoint is to evaluate the induction of adaptive immune responses to the personalized neo-antigen vaccine measured by functional assays and peptide-MHC multimer stainings.

The tertiary objective is to evaluate the clinical efficacy of the treatment. The endpoints will be objective responses (OR), progression free survival (PFS) and overall survival (OS).

DETAILED DESCRIPTION:
Cancer immunotherapy has shown the ability to improve the survival of patients with multiple types of advanced cancers. The human immune system can recognize the products of somatic genetic alterations in tumors, or neo-antigens, which are not expressed on normal cells. These neoantigens are an attractive immune target because their selective expression on tumors can minimize immune tolerance as well as the risk of side effects such as autoimmune reaction.

Although neoantigens are ideal targets for cancer immunotherapies, most neoantigens arise from unique mutations and are not shared between individual patients. Thus, neoantigen-directed immunotherapy will need to be personalized. Novel technical advances in next-generation sequencing allow fast and systematic prediction of cancer neoantigens for each individual patient. Initial attempts of therapeutic cancer vaccination targeting individual neo-antigens have proven non-toxic and met their immunological endpoints.

In this study investigators will use the proprietary platform PIONEER for fast and accurate identification of a neo-antigen vaccine tailored to each individual patient. The vaccine, based on 5-15 peptides derived from a patient's tumor individual neo-antigens, will be formulated with a novel adjuvant to strengthen CD8+ T cell immunity to cancer. Immune checkpoint inhibitors targeting PD-1 or PD-L1 will be administered both before, during and after vaccination to unleash the activity of vaccine-induced immune responses.

ELIGIBILITY:
Inclusion Criteria:

1. Target Disease Exception

   1. The subject must sign and date the IRB/IEC approved written informed consent form prior to the performance of any study-related procedures that are not considered part of standard of care.
   2. Consent for tumor biopsy samples. i. Subject must consent and will be required to undergo a MANDATORY pre-treatment biopsy; therefore, subjects must have a lesion located such that the specimen can be obtained at acceptable clinical risk as judged by the Investigator. The acquisition of existing formalin-fixed paraffin-embedded (FFPE) tumor tissue, either a block or unstained slides, for performance of correlative studies should also be collected if available. Subjects unable to provide a pre-treatment tumor biopsy or do not have accessible lesions are not eligible. If there is only one measurable lesion, and a core-needle biopsy is done (instead of excisional), the lesion may be used as measurable lesion. If there are more than one measurable lesions, the lesion being biopsied should not be a target lesion. Subjects must have histologic or cytologic confirmation of an incurable solid malignancy that is advanced (metastatic and/or unresectable)

      2. Target population

   a) Subjects must have cytologic or histologic confirmation of one of the following selected advanced (metastatic and/or unresectable) solid malignancies: i. Malignant melanoma - Uveal melanoma is NOT eligible ii. Non-small cell lung cancer: squamous or non-squamous histology iii. Bladder carcinoma: transitional cell carcinoma of the urothelium involving the bladder, urethra, ureter, or renal pelvis.

   b) Subjects must fall into one of these two categories: i. Cohort A (limited to max 15 subjects): candidate to treatment with one anti-PD-1 or anti-PD-L1 agent but who had not previously been treated with anti-PD-1 or anti-PD-L1 in the metastatic/unresectable setting.

   ii. Cohort B (limited to max 15 subjects): subjects who are treated continuously for at least 4 months with one anti-PD-1 or anti-PD-L1 agent in the metastatic/unresectable setting, without unequivocal objective response or disease progression, and who qualify for continued treatment with the same agent, who accept a second biopsy.

   c) At least one measurable parameter according to RECIST 1.1.

   d) ECOG performance status of 0 or 1

   e) Life expectancy of >12 weeks at the time of informed consent per Investigator assessment

   f) Adequate organ function as defined by the following hematological and biochemical criteria:

   a. AST and ALT ≤2,5 X ULN or ≤5 X ULN with liver metastases b. Serum total bilirubin ≤1,5 X ULN or direct bilirubin ≤ ULN for patient with total bilirubin level > 1,5 ULN c. Serum creatinine ≤1,5 X ULN d. ANC (Absolute Neutrophil Count) ≥1,000/mcL e. Platelets ≥ 75,000 /mcL f. Hemoglobin ≥ 9 g/dL eller ≥ 5.6 mmol/L

3. Age and reproductive status:

1. Age ≥ 18
2. Women must not be breastfeeding
3. Women of childbearing potential: a negative pregnancy test is mandatory within 72 hours prior to the start of study drug
4. Woman: Agree to use contraceptive methods with a failure rate of < 1 % per year during the treatment period and for at least 150 days after the study treatment. Safe contraceptive methods for women are birth control pills, intrauterine device, contraceptive injection, contraceptive implant, contraceptive patch or contraceptive vaginal ring.
5. Men: if sexually active with women of childbearing potential, agree to use contraceptive measures; agree to refrain from donating sperm

Exclusion Criteria:

1. Target Disease Exception

   a) Subjects with known or suspected CNS metastases or with the CNS as the only site of active disease are excluded with the following exceptions: i. Subjects with controlled brain metastases will be allowed to enroll. Controlled brain metastases are defined as those with no radiographic progression for at least 4 weeks after radiation and/or surgical treatment at the time of consent. Subjects must have been off of steroids for at least 2 weeks prior to informed consent, and have no new or progressive neurological signs and symptoms.
2. Medical History and Concurrent Diseases

   1. Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
   2. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, or carcinoma in situ of the prostate, cervix, or breast.
   3. A known or underlying medical condition that, in the opinion of the Investigator or Sponsor, could make the administration of study drug hazardous to the subject or could adversely affect the ability of the subject to comply with or tolerate study
   4. Requirement for daily supplemental oxygen
   5. The patient has a history of pneumonitis, organ transplant, human immunodeficiency virus positive, active hepatitis B or hepatitis C
   6. Any of the following medications or procedures:

   i. Within 2 weeks prior to time of treatment initiation: I. Systemic or topical corticosteroids at immunosuppressive doses (> 10 mg/day of prednisone or equivalent). Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.

   II. Palliative radiation or gamma knife radiosurgery ii. Within 4 weeks prior to time of treatment initiation: I. Any anticancer drug II. Any vaccine or adjuvant III. Allergen hyposensitization therapy IV. Growth factors V. Major surgery, or the subject has not recovered from surgery at the time of treatment initiation

   g) The subject has not recovered to grade 0-1 from adverse events due to prior chemotherapy, radioactive or biological cancer therapy

   h) History of life-threatening or severe immune related adverse events on treatment with another immunotherapy and is considered to be at risk of not recovering

   i) The subject is expected to require any other form of systemic antineoplastic therapy while receiving the treatment

   j) Any condition that will interfere with patient compliance or safety (including but not limited to psychiatric or substance abuse disorders)

   k) Known, suspected or anticipated side effects to vaccine adjuvants

   l) Significant medical disorder according to investigator; e.g. severe asthma or chronic obstructive lung disease, dysregulated heart disease or dysregulated diabetes mellitus

   m) Concurrent treatment with other experimental drugs

   n) Severe allergy or anaphylactic reactions earlier in life
3. Other exclusion criteria

   1. The patient is unable to voluntarily agree to participate
   2. Prisoners or subjects who are involuntarily incarcerated

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Number and type of reported adverse events | 0-100 weeks
  The primary objective is to assess tolerability and safety of a personalized neo-antigen vaccine containing up to 15 peptides derived from somatic mutation of the individual patient's cancer, with CAF09b as adjuvant. The vaccine formulation will be administered in combination with an approved anti-PD-1 or anti-PD-L1 inhibitor to patients with advanced solid tumors. The endpoint is the characterization of adverse events (AE) assessed by CTCAE 4.0.

SECONDARY OUTCOMES:
Treatment related immune responses | 0-100 weeks
  To evaluate the immunological impact of the treatment. Elispot and tetramer staining methods will be applied to identify NeoPepVac specific T cells in the blood over time

OTHER OUTCOMES:
Overall survival | 3 years
  Overall survival (OS), defined as the time from the start of treatment to death, will be described with the Kaplan-Meier curve.
Objective response rate Progression free survival | 3 years
  Progression-free survival (PFS), defined as the time from start of treatment to disease progression, relapse or death due to any cause, whichever is earlier, will be described with the Kaplan-Meier curve.
Objective response rate | 3 years
  Tumor responses will be evaluated using RECIST1.1 for the assessment of efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Prof., MD, Principal Investigator — CCIT (Center for Cancer Immune Therapy)
Locations (2):
- Denmark (2):
  - Herlev Hospital, Center for Cancer Immune Therapy,, Herlev
  - Herlev Hospital, Herlev

IPD SHARING:
Plan to Share IPD: No